CLINICAL TRIAL: NCT01924299
Title: The Effect of Ketoconazole or Fluconazole on the Pharmacokinetics of Baricitinib in Healthy Subjects
Brief Title: A Study of Baricitinib When Administered With Ketoconazole or Fluconazole in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14607; I4V-MC-JAGJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — baricitinib; Ketoconazole; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baricitinib + Ketoconazole (Experimental): Baricitinib - 10 milligrams (mg) administered orally once on Day 1 of Period 1 and on Day 6 of Period 2.
  Ketoconazole - 400 mg administered orally once daily (QD) for 6 days (Day 3 through Day 8) in Period 2.
  Interventions: Drug: Baricitinib; Drug: Ketoconazole
- Baricitinib + Fluconazole (Experimental): Baricitinib - 10 mg administered orally once on Day 1 of Period 1 and on Day 7 of Period 2.
  Fluconazole - 400 mg administered orally once on Day 3 of Period 2, followed by 200 mg administered orally QD for 6 days (Day 4 through Day 9) in Period 2.
  Interventions: Drug: Baricitinib; Drug: Fluconazole

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
Drug: Ketoconazole — Administered orally
  Arms: Baricitinib + Ketoconazole
Drug: Fluconazole — Administered orally
  Arms: Baricitinib + Fluconazole

SUMMARY:
The main purpose of this study is to look at the effect of ketoconazole and fluconazole on how much baricitinib gets into the blood stream. The study will also look at the tolerability of baricitinib and ketoconazole when given together and the tolerability of baricitinib and fluconazole when given together.

Participants will be recruited into 1 of 2 treatment groups (Group A or Group B). Each treatment group will participate in 2 study periods. Participants will take baricitinib alone in 1 period and baricitinib with either ketoconazole or fluconazole in the other period. This study will last approximately 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy as determined by medical history and physical examination
* Female participants not of childbearing potential due to surgical sterilization (at least 3 months after surgical hysterectomy, bilateral oophorectomy with or without hysterectomy, or bilateral tubal occlusion/ligation) confirmed by medical history or menopause
* Have a body mass index of 18 to 29 kilograms per square meter (kg/m^2), inclusive, at screening

Exclusion Criteria:

* Participants who have previously completed or withdrawn from this study or any other study investigating baricitinib, and have previously received the study drug
* Have known allergies to baricitinib, ketoconazole, fluconazole, related compounds, or any components of the baricitinib, ketoconazole, or fluconazole formulations, or history of significant atopy
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have a current or recent history [less than 30 days prior to screening and/or less than 45 days prior to day of admission to Clinical Research Unit (CRU)] of a clinically significant bacterial, fungal, parasitic, viral (not including rhinopharyngitis), or mycobacterial infection
* Have alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, total bilirubin, or gamma glutamyl transferase (GGT) values above the upper limit of the reference range for the local laboratory at screening or day of admission to CRU
* Have an absolute neutrophil count (ANC) less than 2 times 10^9 per liter (L) [2000 cells per microliter (μL)] at screening or day of admission to CRU. For abnormal values, a single repeat will be allowed
* Intend to use over-the-counter or prescription medication and/or herbal supplements within 14 days prior to dosing and during the study (with the exception of occasional paracetamol, which will be permitted at the discretion of the investigator), or intended use of vitamin supplements from Day 1 until discharge from the CRU
* Have used or intend to use any drugs or substances that are known to be substrates, inhibitors, or inducers of cytochrome P450 (CYP) 3A4, CYP2C9, or CYP2C19 within 30 days prior to dosing and throughout the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, 2-period, fixed-sequence study. Period 1 was from Day 1 through Day 2. Period 2 was from Day 3 through Day 9 for baricitinib + ketoconazole (Group A) and Day 3 through Day 10 for baricitinib + fluconazole (Group B).
Groups:
- Baricitinib + Ketoconazole (Group A): 10 milligrams (mg) baricitinib administered orally once on Day 1 of Period 1 and on Day 6 of Period 2.
  400 mg ketoconazole administered orally once daily (QD) for 6 days (Day 3 through Day 8) in Period 2.
- Baricitinib + Fluconazole (Group B): 10 mg baricitinib administered orally once on Day 1 of Period 1 and on Day 7 of Period 2.
  400 mg fluconazole administered orally once on Day 3 of Period 2, followed by 200 mg administered orally QD for 6 days (Day 4 through Day 9) in Period 2.
Period: Period 1
Arm/Group | Baricitinib + Ketoconazole (Group A) | Baricitinib + Fluconazole (Group B)
Started | 18 | 18
Received Baricitinib | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Baricitinib + Ketoconazole (Group A) | Baricitinib + Fluconazole (Group B)
Started | 18 | 18
Received at Least 1 Dose of Study Drug | 18 | 18
Received Baricitinib | 17 | 17
Completed | 17 | 17
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Baricitinib + Ketoconazole (Group A): 10 mg baricitinib administered orally once on Day 1 of Period 1 and on Day 6 of Period 2.
  400 mg Ketoconazole administered orally QD for 6 days (Day 3 through Day 8) in Period 2.
- Total: Total of all reporting groups
Arm/Group | Baricitinib + Ketoconazole (Group A) | Baricitinib + Fluconazole (Group B) | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (15.0) | 42.7 (13.7) | 42.5 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 16 | 12 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 18 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 16 | 16 | 32
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Plasma Concentration-Time Curve From Time 0 Hour to Infinity [AUC(0-∞)] of Baricitinib Following Single Doses of Baricitinib Alone or Coadministered With Ketoconazole
Time Frame: Days 1 and 6: predose of baricitinib and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hours postdose
Population: All enrolled participants who received study drug (baricitinib in Period 1 and baricitinib + ketoconazole in Period 2) and had PK data to calculate AUC(0-∞) of baricitinib.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Groups:
- Baricitinib (Group A): 10 mg baricitinib administered orally once on Day 1 of Period 1.
- Baricitinib + Ketoconazole (Group A): 10 mg baricitinib administered orally once on Day 6 of Period 2. 400 mg Ketoconazole administered orally QD for 6 days (Day 3 through Day 8) in Period 2.
Arm/Group | Baricitinib (Group A) | Baricitinib + Ketoconazole (Group A)
Number analyzed (Participants) | 18 | 17
nanograms*hour/milliliter (ng*h/mL) | 720 (23) | 868 (24)

2. Primary Outcome: PK: AUC(0-∞) of Baricitinib Following Single Doses of Baricitinib Alone or Coadministered With Fluconazole
Time Frame: Days 1 and 7: predose of baricitinib and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hours postdose
Population: All enrolled participants who received study drug (baricitinib in Period 1 and baricitinib + fluconazole in Period 2) and had PK data to calculate AUC(0-∞) of baricitinib.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Baricitinib (Group B): 10 mg baricitinib administered orally once on Day 1 of Period 1.
- Baricitinib + Fluconazole (Group B): 10 mg baricitinib administered orally once on Day 7 of Period 2. 400 mg fluconazole administered orally once on Day 3 of Period 2, followed by 200 mg administered orally QD for 6 days (Day 4 through Day 9) in Period 2.
Arm/Group | Baricitinib (Group B) | Baricitinib + Fluconazole (Group B)
Number analyzed (Participants) | 18 | 17
ng*h/mL | 698 (24) | 851 (24)

3. Primary Outcome: PK: Maximum Concentration (Cmax) of Baricitinib Following Single Doses of Baricitinib Alone or Coadministered With Ketoconazole
Time Frame: Days 1 and 6: predose of baricitinib and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hours postdose
Population: All enrolled participants who received study drug (baricitinib in Period 1 and baricitinib + ketoconazole in Period 2) and had PK data to calculate Cmax of baricitinib.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Baricitinib (Group A) | Baricitinib + Ketoconazole (Group A)
Number analyzed (Participants) | 18 | 17
nanograms/milliliter (ng/mL) | 106 (27) | 115 (32)

4. Primary Outcome: PK: Cmax of Baricitinib Following Single Doses of Baricitinib Alone or Coadministered With Fluconazole
Time Frame: Days 1 and 7: predose of baricitinib and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hours postdose
Population: All enrolled participants who received study drug (baricitinib in Period 1 and baricitinib + fluconazole in Period 2) and had PK data to calculate Cmax of baricitinib.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Baricitinib (Group B) | Baricitinib + Fluconazole (Group B)
Number analyzed (Participants) | 18 | 17
ng/mL | 103 (36) | 107 (38)

5. Primary Outcome: PK: Time of Maximum Observed Drug Concentration (Tmax) of Baricitinib Following Single Doses of Baricitinib Alone or Coadministered With Ketoconazole
Time Frame: Days 1 and 6: predose of baricitinib and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hours postdose
Population: All enrolled participants who received study drug (baricitinib in Period 1 and baricitinib + ketoconazole in Period 2) and had PK data to calculate Tmax of baricitinib.
Measure: Median (Full Range); unit: hours
Arm/Group | Baricitinib (Group A) | Baricitinib + Ketoconazole (Group A)
Number analyzed (Participants) | 18 | 17
hours | 1.00 [0.50 to 2.00] | 1.00 [0.50 to 2.00]

6. Primary Outcome: PK: Tmax of Baricitinib Following Single Doses of Baricitinib Alone or Coadministered With Fluconazole
Time Frame: Days 1 and 7: predose of baricitinib and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hours postdose
Population: All enrolled participants who received study drug (baricitinib in Period 1 and baricitinib + fluconazole in Period 2) and had PK data to calculate Tmax of baricitinib.
Measure: Median (Full Range); unit: hours
Arm/Group | Baricitinib (Group B) | Baricitinib + Fluconazole (Group B)
Number analyzed (Participants) | 18 | 17
hours | 1.00 [0.50 to 4.00] | 1.00 [0.50 to 3.00]

ADVERSE EVENTS:
Time Frame: Baseline through study completion (up to Day 23).
Groups:
- Baricitinib (Group A); Baricitinib (Group B): 10 mg baricitinib administered orally once on Day 1 of Period 1. Adverse events are reported from baseline through predose on Day 3.
- Ketoconazole (Group A): 400 mg ketoconazole administered orally QD on Day 3 through Day 5 in Period 2. Adverse events are reported from postdose on Day 3 through predose on Day 6.
- Baricitinib + Ketoconazole (Group A): 10 mg baricitinib administered orally once on Day 6 of Period 2. 400 mg ketoconazole administered orally QD on Day 6 through Day 8 in Period 2.
  Adverse events are reported from postdose on Day 6 up to Day 22.
- Fluconazole (Group B): 400 mg fluconazole administered orally once on Day 3 of Period 2, followed by 200 mg administered orally QD on Day 4 through Day 6 in Period 2.
  Adverse events are reported from postdose on Day 3 through predose on Day 7.
- Baricitinib + Fluconazole (Group B): 10 mg baricitinib administered orally once on Day 7 of Period 2. 200 mg fluconazole administered orally QD on Day 7 through Day 9 in Period 2. Adverse events are reported from postdose on Day 7 up to Day 23.
Arm/Group | Baricitinib (Group A) | Ketoconazole (Group A) | Baricitinib + Ketoconazole (Group A) | Baricitinib (Group B) | Fluconazole (Group B) | Baricitinib + Fluconazole (Group B)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/17 | 0/18 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 4/18 | 7/18 | 4/17 | 3/18 | 4/18 | 6/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baricitinib (Group A) (N=18) | Ketoconazole (Group A) (N=18) | Baricitinib + Ketoconazole (Group A) (N=17) | Baricitinib (Group B) (N=18) | Fluconazole (Group B) (N=18) | Baricitinib + Fluconazole (Group B) (N=17)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 6 (7) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days